CLINICAL TRIAL: NCT04451694
Title: Nutritional Follow up After Hospital Discharge for Coronavirus Disease-19
Acronym: NutriCoviDom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI097
Record Dates: First submitted 2020-06-15; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Covid-19
Keywords: nutritional status; malnutrition; diet intervention; sarcopenia; muscle strength
MeSH Terms: conditions — COVID-19; Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 unit outgoing patients: nutritional evaluation and intervention
  Interventions: Other: nutritional intervention

INTERVENTIONS:
Other: nutritional intervention — nutritional evaluation and intervention and orientation towards adapted care establishment

SUMMARY:
Coronavirus infection is responsible for muscle wasting (sarcopenia), especially during prolonged stays in intensive care. Sarcopenia, in its functional aspect also seems major in patients hospitalized for this infection, in non-ICU unit. Weight loss also appears to be significant, despite a prevalence of overweight and obesity in severe forms. Undernutrition in the obese patient is also possible (undernourished obese and sarcopenia obesity). Anosmia and dysgeusia participate in undernutrition by reducing energy intake. The rehabilitation of these patients requires nutritional support (increased protein intake) associated with progressive retraining to physical activity.

An early and proactive management procedure within Coronavirus disease-19 units has been implemented in conjunction with the Transversal Nutrition Unit (TNU). This nutritional care must be continued after discharge. Follow-up by teleconsultation or telephone consultation is put in place after the patient's discharge Primary Objective: Evaluation of nutritional status at the time of admission and discharge and home follow-up in outgoing patients from Coronavirus disease-19 Units Secondary objectives: Description of the evolution of food intake, diversity of food and coverage of needs Evaluation of the muscular strength of the wrist (by grip test in hospital) and on the arms and legs after return home (visual analog scale) Evolution of anosmia and dysgeusia (at the time of hospital admission, at the time of hospital discharge and at home) Level of physical training before infection (IPAQ) Description of the general state of health measured by the performance index - world health organization scale Description of nutritional prescriptions Description of the prevention measures and incidence of Inappropriate Refeeding Syndrome (IRS) Care needs assessments

ELIGIBILITY:
Inclusion Criteria:

* Covid positive (RT-PCR)

Exclusion Criteria:

* Unable to answer questions by telephone or teleconsultation directly or through a relative, minors under 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: complete survey, about 800 patients. No sample List of patients discharged from COVID Units
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
nutritional evaluation | before Covid, at hospital discharge and between 7 and 45 days after discharge
  weight
nutritional evaluation | before Covid, at at the time of hospital admission, at the time of hospital discharge and between 7 and 45 days after discharge
  BMI

SECONDARY OUTCOMES:
muscle strenght | at the time of hospital admission and at the time of hospital discharge
  hand grip
food intake | at the time of hospital admission, at the time of hospital discharge
  Caloric account
food intake | between 7 and 45 days after discharge
  self evaluation of food intake
muscle strenght | between 7 and 45 days after discharge
  self evaluation of muscle strenght
biological nutritional status | at the time of hospital admission, at the time of hospital discharge
  albuminemia transthyretinemia electrolytes dosage inflammation status
anosmia | at the time of hospital admission, at the time of hospital discharge and between 7 and 45 days after discharge
  anosmia and agueusia evolution

CONTACTS AND LOCATIONS:
Locations (1):
- Quilliot, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Treuil M, Mahmutovic M, Di Patrizio P, Nguyen-Thi PL, Quilliot D. Assessment of dynapenia and undernutrition in primary care, a systematic screening study in community medicine. Clin Nutr ESPEN. 2023 Oct;57:561-568. doi: 10.1016/j.clnesp.2023.08.003. Epub 2023 Aug 5. PMID 37739706
- [Derived] Quilliot D, Gerard M, Bonsack O, Malgras A, Vaillant MF, Di Patrizio P, Jaussaud R, Ziegler O, Nguyen-Thi PL. Impact of severe SARS-CoV-2 infection on nutritional status and subjective functional loss in a prospective cohort of COVID-19 survivors. BMJ Open. 2021 Jul 14;11(7):e048948. doi: 10.1136/bmjopen-2021-048948. PMID 34261689